CLINICAL TRIAL: NCT05230329
Title: CME Versus Standard Right Hemicolectomy for Right Sided Cancers
Status: Not yet recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Issam al-Najami, principal investigator, Odense University Hospital
Other Study IDs: IAN012022
Record Dates: First submitted 2022-01-24; First posted 2022-02-08 (Actual); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Colon Cancer
Keywords: complete mesocolic excision; robot; laparoscopic; right sided colon cancer; quality of life
MeSH Terms: conditions — Colonic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Completemesocolic excision by laparoscopy for right sided cancer
  Interventions: Procedure: right sided hemicolectomy, laparoscopy
- Completemesocolic excision by robot for right sided cancer
  Interventions: Procedure: right sided hemicolectomy, laparoscopy
- Standard right hemi colectomy excision by laparoscopy for right sided cancer
  Interventions: Procedure: right sided hemicolectomy, laparoscopy

INTERVENTIONS:
Procedure: right sided hemicolectomy, laparoscopy — Comparison of CME

SUMMARY:
Our aim of this study is to compare the difference in lymph node yield in CME specimens versus those patients having a standard right hemicolectomy for right sided cancer .The secondary aim of this study was to investigate whether there is an interaction between greater lymph node harvest towards increased survival. Another subgroup analysis of this study is to compare the complications and oncological outcome between laparoscopic versus Robotic CME.

Trial Title CME versus standard right hemicolectomy for right sided cancers Internal ref. no. Clinical Phase Trial Design Observational, prospective, international, multi-center study Trial sites 10 sites over 5 different countries Planned Sample Size At least 330 subjects will be enrolled in this study per cohort, including 10% of lost to follow-up patients).

All patients during the enrolment period shall be screened and recorded at sites in order to identify any selection bias Treatment duration 3 years Follow up duration 5 years Planned Trial Period 10 years Objectives Outcome Measures Primary To compare the lymph node yield between complete mesocolic excision versus standard right hemicolectomy for patients with right sided cancer Number of harvested lymph nodes Secondary Incidence of local recurrence after surgery at 2 and 5 years

Disease free survival (2 and 5 years)

5-year overall survival

30-day and 90-day mortality,

60-day postoperative major complications (As measured by the Comprehensive Complication Index (CCI®).)

Pathological quality assessment. Completeness of mesocolon excision (CME) will be assessed by the pathologist

Operative length of time (total OR utilisation time and operative time skin to skin, minutes)

Assessment of intraoperative adverse events within advanced minimally-invasive surgery in order to report "near misses" and associated impact upon clinical outcomes

Conversion to open surgery

For Minimally invasive CME or standard right hemicolectomy - to compare the types of anastomosis (intra-corporeal versus Extra-coporeal ) on anastomosis leak rate 4. 5. 6. 7. Recurrence picked up on intensive follow up schedules with yearly CT scan for 5 years

Definitions:

Distal resected margin ≥ 5cm Lymph node yield Mesocolic plane of surgery Central vascular ligation (within 1cm of ileocolic vessels origins) R0 resection (all margins clear)

Investigational Medicinal Product(s) n/a Formulation, Dose, Route of Administration n/a

DETAILED DESCRIPTION:
CRC is the third most common cancer in men and second most common in women with almost 55% of these cases occurring in more developed nations Findings from a recent population-based study showed that the oncological outcome was worse for right-sided colon cancers than left-sided colon cancers. The authors also noted that the overall survival after curative surgery for right-sided colon cancer was better in patients whose surgery led to a lymph node yield of 22 or more. Other studies also confirmed these findings of better outcome after more extensive lymph node dissection for colon cancer.

To achieve this strategy of increased lymph node yield, a complete mesocolic excision (CME) of the colonic cancer have been proposed. This concept of CME aims to extrapolate the teaching of total mesorectal excision for rectal cancer to colonic cancer by separating the mesocolic from the parietal plane and true central ('high') ligation of the supplying arteries and draining veins. All the lymph nodes along the tumour supplying vessels are contained in the specimen Hohenberger et al have used this technique in 1329 consecutive cases and have found decreased5-year local recurrences rates of colon cancers (from 6.5% to 3.6%) and increased cancer-related 5-year survival rates (82.1% to 89.1%).

However the CME technique remains controversial as the evidence of increased disease-free survival after CME is mainly based on only two single centre studies Complete mesocolic excision is also a more challenging operation than a standard right hemicolectomy. This is due to the complex vascular anatomy of the right colon, and hence many surgeons and surgical units have refrained from performing right-sided complete mesocolic excision.

Nevertheless a few international centres have started to implement CME surgery for right-sided cancers. In Japan for example, central lymph node dissection similar to complete mesocolic excision is recommended for clinical stage T3-4 or pN1-2 tumours. Berthelsen et al recently published their results of central mesocolic lymph node excision on risk of recurrence after resection for right-sided colon adenocarcinoma. They implemented CME as the standard surgical approach for colon cancer in their hospital since 2008.The authors noted that CME has the potential to reduce the risk of recurrence and improve long-term outcome after resection for all UICC stages I-III of right-sided colon adenocarcinomas.

AIM OF THE STUDY Our aim of this study is to compare the difference in lymph node yield in CME specimens versus those patients having a standard right hemicolectomy for right sided cancer .The secondary aim of this study was to investigate whether there is an interaction between greater lymph node harvest towards increased survival. Another subgroup analysis of this study is to compare the complications and oncological outcome between laparoscopic versus Robotic CME.

Right-sided tumours is defined as any primary adenocarcinoma located in the caecum, the ascending colon, the hepatic flexure, and the right or mid-third of the transverse colon

Minimal invasive operative techniques for CME and Standard right hemicolectomy CME has been performed via laparotomy for many years. Minimal access colorectal surgery has matured steadily over the last decades hence there have been questions asked whether CME can be performed safely and adequately using minimal access techniques.

Continuous progress in technology [application of high-definition (HD) and three-dimensional (3D) and other camera systems, has led to claims of improved precision in lymph node dissection and vascular sceletonization.

Several studies have now reported that laparoscopic CME resection was feasible and did not compromise patient safety. However theses studies were from single institution and were non-comparative small studies.

Robotic right hemicolectomy (RRHC) has been subject to much interest in recent years from its potential dual learning benefits to the operating colorectal surgeon and clinical benefits to the patients. The potential benefits of robotic systems over conventional laparoscopy include superior three-dimensional vision, seven degrees of freedom of movement replicating the surgeon's hand movements, lack of tremor and potential superior ergonomics, suggesting potential application in both routine and more difficult cases Currently there is little if any literature specifically comparing laparoscopic to robotic CME. Hence we also aim to compare the complications and oncological outcome between laparoscopic versus Robotic versus open CME Intra-corporeal anastomosis Formation With minimally invasive surgery for CME and standard right hemicolectomy there have been an increase in intra-corporeal anastomosis formation. The increased dexterity, third-hand retraction and better visualization at Robotic right hemicolectomy can allow for less colonic dissection, less disturbance of the natural embryological lie of tissue planes, elimination of traction and possible twisting on the remaining transverse colon.

Several studies have revealed conflicting results with some showing significantly fewer conversions for the minimally invasive surgery intra-corporeal anastomosis when compared to the extracorporeal approach and others that show no significant difference.

Hence we aim to do a subset analysis on the anastomotic leak rate between the robotic intra-corporeal anastomosis versus laparoscopic intra-corporeal anastomosis versus minimally invasive surgery extra-corporeal anastomosis.

Anastomosis leak will be defined as sepsis in the post operative period with raised inflammatory markers requiring antibiotics or CT scan confirming free gas around anastomosis or patient return to theatre showing anastomosis breakdown intraoperatively

It will be up to the individual surgeon as to the preferred method of anastomosis they use for each case

5. OBJECTIVES AND OUTCOME MEASURES Objectives Outcome Measures Timepoint(s) of evaluation of this outcome measure (if applicable) Primary Objective The primary aim of the study is to compare the lymph node yield between CME and standard right hemicolectomy in right sided cancers Number of harvested lymph nodes Within 30 days of operation Secondary Objectives Surgical morbidity/mortality up to 90 days

Pathological quality assessment

Incidence of local recurrence after surgery at 2 and 5 years

Overall survival at 5 and 10 years

Assessment of intraoperative adverse events of the surgery

Health economics assessements

Conversion to open surgery

Evaluation of the operative length of time

For Minimally invasive CME or standard right hemicolectomy - to compare the types of anastomosis (intra-corporeal versus Extra-coporeal )

Completeness of CME will be assessed by the pathologist and is defined as:

* Distal resected margin ≥ 5cm
* Lymph node yield
* Mesocolic plane of surgery
* Central vascular ligation (within 1cm of ileocolic vessels origins)
* R0 resection (all margins clear) Local recurrence is defined according to first documented clinical or imaging relapse or the date of death from any cause, whichever occurs first.

To report "near misses" and associated impact upon clinical outcomes

Healthcare resource utilization (costs) including hospital length of stay, ICU hours.

Total OR utilisation time and operative time skin to skin, minutes

Anastomosis leak rate

At 30 and 60 days after surgery

LR is defined as the interval from date of randomisation to the date of first evidence of disease progression wholly within the colon and/or distally. Distant failure or death will be considered as a competing risk.

Defined as sepsis with raised inflammatory markers requiring antibiotics or CT scan confirmed free gas around anastomosis or patient return to theatre showing anastomosis breakdown intraoperatively

6. TRIAL DESIGN This is an observational prospective, multicentre trial Patients will be having either a minimally invasive (laparoscopic/Robotic) CME versus a standard minimally invasive right hemicolectomy ( laparoscopic/Robotic ) for right sided cancers.

Right-sided tumours is defined as any primary adenocarcinoma located in the caecum, the ascending colon, the hepatic flexure, and the right or mid-third of the transverse colon Distal Transverse colon and splenic flexure tumors will be excluded to minimize misclassification bias The study will include 330 patients from UK and a number of international sites including, but not limited to, Denmark, Germany, Japan , The Netherlands and Australia This study has no impact on staging investigations, timing of surgery or any other aspect of the patients' pre, peri or post-operative care.

All decisions remain with the local clinician multi-disciplinary team including when to discharge from hospital.

7. PARTICIPANT IDENTIFICATION 7.1. Trial Participants Participants with right sided cancer who are scheduled for initial treatment by either CME or standard right hemicolectomy 7.2. Inclusion Criteria

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Undergoing CME or standard right hemicolectomy surgery for right-sided cancer after MDT discussion.
* Cancer must be confirmed by histological, radiological, endoscopic diagnosis
* In the Investigator's opinion, is able and willing to comply with all trial requirements.
* Willing to allow his or her General Practitioner and consultant, if appropriate, to be notified of participation in the trial.

7.3. Exclusion Criteria

The participant may not enter the trial if ANY of the following apply:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Participant with life expectancy of less than 6 months.
* Distal Transverse colon and splenic flexure tumors
* Evidence of T4 disease invading adjacent organs
* Synchronous surgical procedure planned with CME or right hemicolectomy
* Urgent, unplanned or emergency surgery
* Neoadjuvant chemotherapy administered to treat this cancer prior to resection
* Concurrent or previous abdominal or pelvic malignancy within five years prior to registration irrespective of treatment modality
* Known Crohn's disease with active terminal ileal disease
* Evidence of systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude surgery, or other severe incapacitating disease, i.e. ASA IV (a patient with severe systemic disease that is a constant threat to life) or ASA V (a moribund patient who is not expected to survive without the operation).
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

  8. TRIAL PROCEDURES 8.1. Recruitment Patients undergoing either CME surgery or standard right hemicolectomy for right sided cancer will be given information about the trial around the time of surgery planning outpatient clinic visit. Patients will be discussed in the weekly colorectal MDT meeting prior to eligibility assessment. Suitable patients will be identified at this stage. Patients will then be approached, screened and recruited in the colorectal outpatient clinic at the routine pre-operative visit.

8.1. Screening and Eligibility Assessment Patient screening and eligibility will be determined at the routine pre-operative clinic visit. No special screening procedures are required.

Informed Consent The participant must personally sign and date the latest approved version of the Informed Consent form before any trial specific procedures are performed.

Written and verbal versions of the Participant Information and Informed Consent will be presented to the participants detailing no less than: the exact nature of the trial; what it will involve for the participant; the implications and constraints of the protocol; the known side effects and any risks involved in taking part. It will be clearly stated that the participant is free to withdraw from the trial at any time for any reason without prejudice to future care, without affecting their legal rights and with no obligation to give the reason for withdrawal.

The participant will be allowed as much time as wished to consider the information, and the opportunity to question the Investigator, their GP or other independent parties to decide whether they will participate in the trial. Written Informed Consent will then be obtained by means of participant dated signature and dated signature of the person who presented and obtained the Informed Consent. The person who obtained the consent must be suitably qualified and experienced, and have been authorised to do so by the Chief/Principal Investigator. A copy of the signed Informed Consent will be given to the participant. The original signed form will be retained at the trial site.

8.2. Baseline Assessments Baseline assessments will include the histopathology of the cancer biopsied, and CEA level

Subsequent Visits These visits are all part of the standard clinical care following CME or standard right hemicolectomy surgery for right-sided cancer, so no extra visits are involved.

The following assessments are required for this study to assess disease recurrence up to 5 years.

* Colonoscopy (or CT Colonography) at 60 months post surgery
* CT- Chest, Abdo, Pelvis 1 and 3 years post surgery

8.3. Discontinuation/Withdrawal of Participants from Trial Treatment

Each participant has the right to withdraw from the trial at any time. In addition, the Investigator may discontinue a participant from the trial at any time if the Investigator considers it necessary for any reason including:

* Pregnancy
* Ineligibility (either arising during the trial or retrospectively having been overlooked at screening)
* Significant protocol deviation
* Significant non-compliance with treatment regimen or trial requirements
* Withdrawal of Consent
* Loss to follow up Patients who withdraw from the trial will continue to be offered surveillance as part of routine follow up after right colon cancer treatment. Data collected on patients who withdraw from the trial will be analysed according to intention-to-treat.

The reason for withdrawal will be recorded in the CRF. If the participant is withdrawn due to an adverse event, the Investigator will arrange for follow-up visits or telephone calls until the adverse event has resolved or stabilised.

8.4. Definition of End of Trial The end of trial is the date of the last follow up of the last participant.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.
* Male or Female, aged 18 years or above.
* Undergoing CME or standard right hemicolectomy surgery for right-sided cancer after MDT discussion.
* Cancer must be confirmed by histological, radiological, endoscopic diagnosis
* In the Investigator's opinion, is able and willing to comply with all trial requirements.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the trial.
* Participant with life expectancy of less than 6 months.
* Distal Transverse colon and splenic flexure tumors
* Evidence of T4 disease invading adjacent organs
* Synchronous surgical procedure planned with CME or right hemicolectomy
* Urgent, unplanned or emergency surgery
* Neoadjuvant chemotherapy administered to treat this cancer prior to resection
* Concurrent or previous abdominal or pelvic malignancy within five years prior to registration irrespective of treatment modality
* Known Crohn's disease with active terminal ileal disease
* Evidence of systemic disease (cardiovascular, renal, hepatic, etc.) that would preclude surgery, or other severe incapacitating disease, i.e. ASA IV (a patient with severe systemic disease that is a constant threat to life) or ASA V (a moribund patient who is not expected to survive without the operation).
* Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the trial, or may influence the result of the trial, or the participant's ability to participate in the trial.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants with right sided cancer who are scheduled for initial treatment by either CME or standard right hemicolectomy
Sampling Method: Probability Sample
Enrollment: 330 (Estimated)
Dates: Start 2022-03-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2028-02-01 (Estimated)

PRIMARY OUTCOMES:
we will assess the Number of harvested lymph nodes after colonic resectio | 3 years anticipated
  The primary aim of the study is to compare the lymph node yield between CME and standard right hemicolectomy in right sided cancers

SECONDARY OUTCOMES:
mortality and morbidity | 90 days
  Surgical morbidity/mortality up to 90 days compared in the three groups
Pathological quality assessment | 90 days
  Completeness of CME will be assessed by the pathologist and is defined as:
  * Distal resected margin ≥ 5cm
  * Lymph node yield
  * Mesocolic plane of surgery
  * Central vascular ligation (within 1cm of ileocolic vessels origins)
  * R0 resection (all margins clear)
Incidence of local recurrence after surgery at 1,3 and 5 years | 5 years
  Local recurrence is defined according to first documented clinical or imaging relapse or the date of death from any cause, whichever occurs first.
  LR is defined as the interval from date of randomisation to the date of first evidence of disease progression wholly within the colon and/or distally. Distant failure or death will be considered as a competing risk.
Overall survival at 5 and 10 years | 10 years
  Overall survival at 5 and 10 years
Assessment of intraoperative adverse events of the surgery | 90 days
  To report "near misses" and associated impact upon clinical outcomes Conversion to open surgery
  Evaluation of the operative length of time
  For Minimally invasive CME or standard right hemicolectomy - to compare the types of anastomosis (intra-corporeal versus Extra-coporeal ) Anastomosis leak rate Defined as sepsis with raised inflammatory markers requiring antibiotics or CT scan confirmed free gas around anastomosis or patient return to theatre showing anastomosis breakdown intraoperatively.
Health economics assessements | 24 months
  Healthcare resource utilization (costs)
Health related quality of life | 1, 3 and 5 years
  Validated eortc qlq c-29.
Health related quality of life | 1,3 and 5 years
  eortc qlq c-30
Health related quality of life | 1,3 and 5 years
  euroqol eq-5d

CONTACTS AND LOCATIONS:
Overall Officials: Issam Al-Najami, M.D Ph.D., Principal Investigator — Odense University hospital, department of colorectal surgery
Locations (1):
- Issam al-Najami, Svendborg, Southern Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No